CLINICAL TRIAL: NCT02893228
Title: Does Saline Injection Around Phrenic Nerve Reduce Incidence of Diaphragmatic Paresis Following Interscalene Block?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Adelaide and Meath Hospital, incorporating The National Children's Hospital (Other)
Responsible Party: Principal Investigator, Karthikeyan Kallidaikurichi Srinivasan, Doctor, The Adelaide and Meath Hospital, incorporating The National Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AMNCH-A-SIPPIB
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Phrenic Nerve Palsy
Keywords: forced expiratory volume in 1 second; forced vital capacity; peak expiratory flow rate; interscalene block; diaphragmatic paresis
MeSH Terms: interventions — Sodium Chloride; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (saline group) (Experimental): In plane posterior approach will be used with a 50mm short bevel block needle (Braun), advanced through the middle scalene muscle. At the location chosen for interscalene block the needle tip will be positioned anterior to the anterior scalene muscle. At this point 10ml of 0.9% saline will be injected. This will be followed by repositioning of the needle between roots C5 and C6 where 20 ml of 0.25% levobupivicaine will be injected in 5ml increments with intermittent aspiration.
  Interventions: Procedure: Saline; Drug: Levobupivacaine
- Group C (control group) (Active Comparator): In plane posterior approach will be used with a 50mm short bevel block needle (Braun), advanced through the middle scalene muscle. The needle tip will be positioned between roots C5 and C6 where 20 ml of 0.25% levobupivicaine will be injected in 5ml increments with intermittent aspiration.
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Procedure: Saline — At the location chosen for interscalene block the needle tip will be positioned anterior to the anterior scalene muscle. At this point 10ml of 0.9% saline will be injected.
  Arms: Group S (saline group)
Drug: Levobupivacaine — the needle tip will then be positioned between C5 and C6 nerve roots. At this location, 20 ml of 0.25% levobupivacaine will be injected in 5 ml increments with intermittent aspiration. The needle tip will not be repositioned unless the patient complaints of paraesthesia

SUMMARY:
Hemi-diaphragmatic palsy is a common undesirable effect of interscalene block, with an incidence of up to 100%. Mechanism of palsy is thought to be related to spread of local anaesthetic anterior to the anterior scalene muscle. We hypothesize that by injecting saline in this anatomical location prior to performing an interscalene block the incidence of phrenic palsy will be reduced.

DETAILED DESCRIPTION:
Patients will be randomised to either group S (saline group) or group C (conventional group) by computer generated random numbers and allocation will be enclosed in sealed envelope. Anaesthetist performing and/or supervising the block will be the only personnel who will be aware of the randomisation. Patients will be blinded to the study group. Intraoperative management of the case will be done by an anaesthetist blinded to the study group. Outcome measurements will be recorded by study observers blinded to the group allocation.

ISB protocol Following written informed consent, the patient will have routine monitors attached (ECG, Pulse oximeter and non-invasive blood pressure). Intravenous access will be secured and patients will be placed in 45 degree head-up position for the block with head turned to the non-operative side. Intravenous sedation with Midazolam (2 mg) and fentanyl (50 to 100 microgram) will be administered to all patients prior to the block. The ultrasound machine will be positioned on the side opposite to the block. Skin will be prepped with 2% Chlorhexidine (Chloraprep) following which the block will be performed under strict aseptic precautions with the anesthetist wearing a mask and sterile gloves. The high frequency linear probe (sonosite) will be aligned transversely across the neck at the interscalene level to identify C5 and C6 nerve roots. 2% lidocaine will be used for skin infiltration and "stop before block" performed prior to insertion of block needle. In plane posterior approach will be used with a 50 mm short bevel block needle (Braun) advanced through middle scalene muscle. Following this, the technique differs between the two groups.

In group C, the needle tip will then be positioned between C5 and C6 nerve roots. At this location, 15 ml of 0.25% levobupivacaine will be injected in 5 ml increments with intermittent aspiration. The needle tip will not be repositioned unless the patient complaints of paraesthesia.

In group S, at the same level chosen for interscalene block, needle tip will be positioned anterior to anterior scalene muscle. At this location 10 ml 0.9% saline will be injected. This will then be followed by repositioning of needle between roots of C5 and C6 where 15 ml of 0.25% levobupivacaine will be injected in 5 ml increments with intermittent aspiration. The needle tip will not be repositioned unless the patient complaints of paraesthesia.

Intra-operative procedure

Following performance of the block, all patients will receive protocolised general anaesthetic. Anaesthesia will be induced with 2-3 mg per kg of propofol, followed by rocuronium 0.6mg/kg for muscle relaxation. Anaesthesia will be maintained with inhaled sevoflurane (MAC 1 end tidal concentration) along with air and oxygen mixture to deliver an inspired oxygen concentration of 40%. Antibiotics will be given as per hospital protocol prior to incision. In the absence of contraindications, all patients will receive intravenous paracetamol 1g and parecoxib 40 mg as a part of multimodal analgesia regimen. All patients will also receive intravenous dexamethasone 8 mg and ondansetron 4mg for post-operative nausea and vomiting prophylaxis. Further doses of fentanyl in 25 microgram increments will be administered by the anaesthetist if the heart rate increases by more than 15% of baseline values obtained prior to induction. Patients will be reversed by suggamadex. If at least two twitches are present during TOF measurement 2 mg/kg dose will be administered. If less than 2 twitches are present, 4 mg/kg dose will be administered.

Post-operative procedure:

Following transfer to recovery unit, if patient reported pain score by numerical rating score was >3, morphine 2 mg increments will be given intravenously by the recovery staff. This will be repeated every 5 minutes till the pain score is <4. In patients needing more than 10 mg of morphine in the recovery, anaesthetist will be requested to review the patient. Post-operatively, in the absence of contraindications, all patients will be prescribed regular paracetamol 1g, 6 hourly and celecoxib 200 mg, 12 hourly. For breakthrough pain, oxynorm 10 mg as needed once every 4 hours will be prescribed. Anti-emetics (ondansetron 4 mg, 8 hourly and Cyclizine 50 mg, 8 hourly) will be prescribed for all patients to be administered as required. Patient will also be asked about presence or absence of subjective feeling of dypnoea and report satisfaction of overall anaesthetic management (numerical rating scale 0-10) prior to discharge from recovery.

Diaphragm palsy and PFT assessment Diaphragm assessment and bed side spirometry will be done at two time points. First measurement (time point 1) will be done at the baseline as soon as the patient arrives in the induction room. This will be done prior to administration of any sedative agents or regional block. Second assessment (time point 2) will be done post-operatively once the patients are deemed to be ready for discharge from recovery back to the ward.

For diaphragmatic paresis assessment, patients will be placed in supine position and curvilinear ultrasound probe (2-5 MHz) will be used. Diaphragm will be identified as hyperechoic line by subcostal approach using liver and spleen as acoustic windows. Patients will be requested to take deep breaths and M mode will be used to measure the excursion of diaphragm. Diaphragmatic paresis will be documented when there is more than 75% reduction in the excursion compared to baseline or if there was paradoxical movement of the diapragm. Bedside assessment will be done by radiologist blinded to the study group.

Bedside spirometry assessments will be done with patients sitting up. They will be requested to make maximum inspiratory effort and blow as hard and fast in to the device. Best reading from three repeated measurements will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery on shoulder, humerus, or clavicle

Exclusion Criteria:

* Patient refusal
* Allergy to local anaesthesia
* Severe coagulopathy
* Contralateral phrenic nerve palsy
* Local infection
* Moderate to severe pulmonary dysfunction (GOLD II, II, IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Rate of diaphragmatic paresis recorded in the post-operative period identified by ultrasound assessment | 4 hours
  Diaphragmatic paresis will be documented with greater than 75% reduction in excursion compared to baseline

SECONDARY OUTCOMES:
FEV1 | 4 hours
  Forced expiratory volume in 1 second (FEV1)
FVC | 4 hours
  Forced vital capacity (FVC)
PEFR | 4 hours
  Peak expiratory flow rate (PEFR) will be assessed and compared to baseline
Pain control | 24 hours post-opertive
  Intra-operative fentanyl consumption, post-operative morphine consumption in 24 hours, pain scores (numerical 1-10) on arrival in recovery and at 24 hours post operatively

OTHER OUTCOMES:
Patient satisfaction | 4 hours
  Patient satisfaction scores obtained prior to discharge from recovery will be obtained by numerical rating score 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Srinivasan, MD., FCARCSI, Principal Investigator — Adelaide and Meathe Hospital, Incorporating National Children's Hospital
Locations (1):
- Adelaide and Meath Hospital, Incorporating National Children Hospital, Tallagh, Dublin 24, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Urmey WF, Grossi P, Sharrock NE, Stanton J, Gloeggler PJ. Digital pressure during interscalene block is clinically ineffective in preventing anesthetic spread to the cervical plexus. Anesth Analg. 1996 Aug;83(2):366-70. doi: 10.1097/00000539-199608000-00028. PMID 8694320
- [Background] Urmey WF, McDonald M. Hemidiaphragmatic paresis during interscalene brachial plexus block: effects on pulmonary function and chest wall mechanics. Anesth Analg. 1992 Mar;74(3):352-7. doi: 10.1213/00000539-199203000-00006. PMID 1539813
- [Background] Cangiani LH, Rezende LA, Giancoli Neto A. Phrenic nerve block after interscalene brachial plexus block. Case report. Rev Bras Anestesiol. 2008 Mar-Apr;58(2):152-9. doi: 10.1590/s0034-70942008000200007. English, Portuguese. PMID 19378533
- [Background] Rau RH, Chan YL, Chuang HI, Cheng CR, Wong KL, Wu KH, Wei TT. Dyspnea resulting from phrenic nerve paralysis after interscalene brachial plexus block in an obese male--a case report. Acta Anaesthesiol Sin. 1997 Jun;35(2):113-8. PMID 9293653
- [Background] Wennike N, Thompson A. Interscalene block as a precipitant of respiratory dysfunction. Br J Hosp Med (Lond). 2012 Apr;73(4):227. doi: 10.12968/hmed.2012.73.4.227. No abstract available. PMID 22585200
- [Background] Sinha SK, Abrams JH, Barnett JT, Muller JG, Lahiri B, Bernstein BA, Weller RS. Decreasing the local anesthetic volume from 20 to 10 mL for ultrasound-guided interscalene block at the cricoid level does not reduce the incidence of hemidiaphragmatic paresis. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):17-20. doi: 10.1097/aap.0b013e3182030648. PMID 21751435
- [Background] Lee JH, Cho SH, Kim SH, Chae WS, Jin HC, Lee JS, Kim YI. Ropivacaine for ultrasound-guided interscalene block: 5 mL provides similar analgesia but less phrenic nerve paralysis than 10 mL. Can J Anaesth. 2011 Nov;58(11):1001-6. doi: 10.1007/s12630-011-9568-5. Epub 2011 Aug 20. PMID 21858614
- [Background] Palhais N, Brull R, Kern C, Jacot-Guillarmod A, Charmoy A, Farron A, Albrecht E. Extrafascial injection for interscalene brachial plexus block reduces respiratory complications compared with a conventional intrafascial injection: a randomized, controlled, double-blind trial. Br J Anaesth. 2016 Apr;116(4):531-7. doi: 10.1093/bja/aew028. PMID 26994230
- [Background] Stundner O, Meissnitzer M, Brummett CM, Moser S, Forstner R, Kokofer A, Danninger T, Gerner P, Kirchmair L, Fritsch G. Comparison of tissue distribution, phrenic nerve involvement, and epidural spread in standard- vs low-volume ultrasound-guided interscalene plexus block using contrast magnetic resonance imaging: a randomized, controlled trial. Br J Anaesth. 2016 Mar;116(3):405-12. doi: 10.1093/bja/aev550. PMID 26865133